CLINICAL TRIAL: NCT04396405
Title: Investigation of Factors Affecting Cardiorespiratory Fitness in Individuals With Systemic Hypertension
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ebru Calik Kutukcu, Associate professor, Hacettepe University
Other Study IDs: GO 20/360
Record Dates: First submitted 2020-05-08; First posted 2020-05-20 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Systemic Hypertension; Muscle Weakness; Vascular Stiffness
MeSH Terms: conditions — Hypertension; Muscle Weakness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to investigate the factors affecting cardiorespiratory fitness in individuals with systemic hypertension.

DETAILED DESCRIPTION:
Systemic artery hypertension is a condition characterized by persistent high blood pressure (BP) in systemic arteries. Blood pressure is expressed as the rate of systolic BP (SBP) (pressure exerted by the blood on the arterial walls when the heart contracts) and diastolic BP (DBP) (pressure that occurs when the heart is relaxed).

Hypertension is defined as SBP level ≥ 140 mmHg and DBP level ≥ 90 mmHg. Pre-hypertension, defined as the gray area, or increased normal blood pressure, ranges between SBP 130-139 mmHg and DBP 85-89 mmHg. Hypertension is among the most common preventable risk factors for cardiovascular diseases. Although hypertension, which is seen as a silent killer due to the absence of any symptoms in its early stages until a serious medical crisis such as heart attack, stroke or chronic kidney disease, is often asymptomatic, some patients may present with headache, dizziness, visual impairment or fainting spells. There is still too much uncertainty about the pathophysiology of hypertension. Fewer patients (between 2% to 5%) as the cause of increased blood pressure; there is an underlying kidney or adrenal disease. However, one reason is not clearly defined and in the rest condition "essential hypertension" is defined. A number of physiological mechanisms are involved in maintaining normal blood pressure, and irregularities of these mechanisms play a role in the development of essential hypertension. These physiological mechanisms; cardiac output and peripheral resistance, renin-angiotensin-aldosterone system, autonomic nervous system, vasoactive substances, excessive coagulation, insulin sensitivity, genetic factors, diastolic dysfunction and endothelial dysfunction.

Evaluation of exercise capacity and prescribing individualized exercise programs in individuals with increased cardiovascular risk and risk factors is a protective and therapeutic health policy. Hypertensive individuals should be evaluated to evaluate motor and cardiovascular functions and prescribe exercise. Hypertension and the chronic diseases it may cause make it difficult for individuals to perform their daily life activities and may limit the participation of individuals in daily life. The exercise, being one of the most important components involved in the management of hypertension together hypertensive subjects of exercise capacity, activities of daily living (ADL), is considerably less than the studies that assessed in detail the balance parameters and the impact of hypertension as it is made in almost all geriatric population of the studies makes it difficult to demonstrate directly. The aim of our study is to evaluate individuals in terms of all these variables and to determine the factors affecting them, to examine the effect of antihypertensive drugs on daily life activity and exercise capacity, and to examine whether gender differences are observed.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or older,
* Having been diagnosed with primary or secondary hypertension,
* Volunteering to participate in the study,

Exclusion Criteria:

* Has a neurological, cognitive or orthopedic disease that will affect the measurements, Having severe respiratory disease (FEV1 <35%; FVC <50%),
* Presence of acute infection,
* Malignancy
* Dementia,
* Having hormone replacement therapy,
* Have had any cardiovascular events in the last 6 months,
* Body mass index is more than 40 kg / cm2,
* Ejection fraction less than 50%,
* Uncontrolled hypertension, diabetes,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable hypertension patients between the ages of 18-65, who are in accordance with the criteria for inclusion in the clinical condition of Hacettepe University Faculty of Medicine, Department of Cardiology and Department of Nephrology from Hacettepe University Faculty of Medicine, Department of Internal Diseases, are included in the study. and who reffered to the Cardiopulmonary Rehabilitation Unit for Physiotherapy also who are willing to participate in the study will be include in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 1 year
  Exercise capacity assesment with six minute stepper test
Submaximal Exercise Capacity | 1 year
  Exercise capacity assesment with six minute walk test

SECONDARY OUTCOMES:
Quality of Life assesment | 1 year
  Quality of Life assesment with Short form 36
Arterial Stiffness | 1 year
  Pulse wave variability
Medication Adherence | 1 year
  Hill Bone Medication Adherence
Physical Activity | 1 year
  Physical Activity assessed with IPAQ
Ventricular functions ve ventricular structure | 1 year
  Left and right ventricular function assessed with ecocardiography

CONTACTS AND LOCATIONS:
Overall Officials: EBRU CALIK-KUTUKCU, PhD, Principal Investigator — Hacettepe University; LALE TOKGOZOGLU, MD, Study Chair — Hacettepe University; YUSUF ZIYA SENER, MD, Study Chair — Hacettepe University; TOLGA YILDIRIM, MD, Study Chair — Hacettepe University; JABRAYİL JABRAYİLOV, MD, Study Chair — Hacettepe University; BEYZA NUR KARADUZ, MsC, Study Chair — Hacettepe University; BURCU OZCAN, MsC, Study Chair — Hacettepe University; DENİZ INAL-INCE, PhD, Study Chair — Hacettepe University; MELDA SAGLAM, PhD, Study Chair — Hacettepe University; NACİYE VARDAR-YAGLI, PhD, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No